CLINICAL TRIAL: NCT02996279
Title: Impact of Chorioamnionitis on Maternal and Fetal Levels of Proinflammatory S100A12
Brief Title: Chorioamnionitis and Proinflammatory S100A12
Acronym: S100A12
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, MARIA PIA DE CAROLIS, MD, Catholic University of the Sacred Heart
Other Study IDs: 100093
Record Dates: First submitted 2016-11-25; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Chorioamnionitis Affecting Fetus or Newborn
Keywords: Neonate; Chorioamnionitis; S100A12
MeSH Terms: conditions — Chorioamnionitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — MATERNAL, CORD AND NEONATAL BLOOD
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- group 1: maternal chorioamnionitis
- group 2: no maternal chorioamnionitis

SUMMARY:
Histologic chorioamnionitis (HCA) may lead to the fetal inflammatory response syndrome (FIRS) and increased levels of proinflammatory molecules.

DETAILED DESCRIPTION:
Histologic chorioamnionitis (HCA) may lead to the fetal inflammatory response syndrome (FIRS). The aim of this pilot study was to evaluate S100A12, a marker of innate immune activation, in mothers with or without HCA and in their infants.

Concentrations of S100A12, Interleukin 6 (IL-6) and C-reactive protein (CRP) were evaluated in maternal, cord, and neonatal blood of very preterm infants. Histologic examinations of placentae and umbilical cords were performed.

ELIGIBILITY:
Inclusion Criteria:

Preterm Birth

Exclusion Criteria:

Congenital Abnormalities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Very Premature Mother-Neonate Pairs
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
S100A12 in Presence of Maternal Chorioamnionitis | 1 Year
  Levels of S100A12 in Maternal, Cord and Neonatal Blood in the Presence or Absence of HCA

IPD SHARING:
Plan to Share IPD: No